CLINICAL TRIAL: NCT06593145
Title: Application of the Autologous CAR T Cells (Tarcidomgen Kimleucel) in the Treatment of Refractory and Relapsed CD19+ B Cell Neoplasms
Brief Title: CAR T Cells in the Treatment of Refractory and Relapsed CD19+ B Cell Neoplasms
Acronym: CARLA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: FamiCordTx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-005720-37
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Mantle Cell Lymphoma (MCL); Large B-cell Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FCTX-CL19-1 (Tarcidomgen Kimleucel) (Experimental): FCTX-CL19-1 (Tarcidomgen Kimleucel) - active IMP - consists of autologous T-cells with chimeric antigen receptor (CAR), Advanced Therapy Medicinal Product, ATMP, Gene Therapy Medicinal Product, GTMP
  Interventions: Biological: FCTX-CL19-1 (Tarcidomgen Kimleucel)

INTERVENTIONS:
Biological: FCTX-CL19-1 (Tarcidomgen Kimleucel) — It will be administered only by Investigators during hospitalization. Each patient will receive one administration of IMP on Day 0:
  * administration route - intravenous
  * cell dose: 0,2 x 106 -2 x 106 CAR T cells per kilogram of patient body weight

SUMMARY:
One arm, open label study to assess the clinical use of Investigational Medicinal Product FCTX-CL19-1 (scientific name: Tarcidomgen Kimleucel) containing autologous anti-CD19 CAR T cells with a preliminary determination of the safety of intravenous IMP administration in patients diagnosed with refractory and relapsed CD19 + B cell neoplasms.

DETAILED DESCRIPTION:
The aim of the study is to determine the safety of therapy with the study medicinal product FCTX-CL19-1 (Tarcidomgen Kimleucel) with preliminary determination of efficacy, as part of a phase I clinical trial in patients with relapsed and refractory B-cell CD19+ tumors.

The hypothesis of the study assumes that the use of the newly developed product FCTX-CL19-1 (Tarcidomgen Kimleucel) containing autologous anti-CD19 CAR T cells is safe and will lead to remission of B-cell cancer resistant to current treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18-65 both inclusive;
2. Diagnosis of:

   1. Refractory B-ALL (acute lymphocytic leukemia) - relapse after hematopoietic cell transplantation, second or more relapse in patients when transplantation is contraindicated)
   2. Large B-cell lymphoma including DLBCL NOS, lymphoma with high level of malignancy, follicular lymphoma transformed to DLBCL and primary mediastinal lymphoma - refractory or relapse or after at least 2 lines of systemic treatment)
   3. Mantle cell lymphoma (MCL) - relapsing or refractory after at least 2 lines of systemic treatment; Diagnostics of individual diagnoses (criteria for complete remission and partial responses for individual disease entities) was developed on the basis of current (July 2022) recommendations of experts of the Polish Society of Clinical Oncology
3. Confirmed CD19 expression on malignant cells;
4. General condition measured by ECOG (Eastern Cooperative Oncology Group) ≤ 1;
5. Patient's weight between 40 kg - 130 kg
6. Sufficient general condition of organs on screening visit:

   1. ALT/AST <2,5 of UNL and bilirubin <1,5 mg/dl (<4 mg/dl for patients with Gilbert syndrome)
   2. Ejection fraction (EF) >50% confirmed in ECHO with no signs of exudation in pericardium during 6 weeks before screening
   3. Saturation of arterial blood >93% with no oxygen insufflation, with no significant exudation in pleural cavity
   4. Serum creatinine clearance >60 ml/min (by Cockcroft-Gault formula);
7. Negative result for HCV, HBV, HIV, Syphilis;
8. Negative test for pregnancy (serum or urine) in the screening visit and/or 7 days before leucapheresis and 7 days before lymphodepleting therapy in women in reproductive age;
9. Assumption of at least 12 months of survival time from screening visit;
10. Agreement to maintain sufficient method of contraception from the date of signing informed consent to 6 months after CART therapy;
11. The last dose of SARS-CoV-2 vaccination taken at least 6 months prior to study enrollment
12. Capable of providing written informed consent;
13. Patients polish native language speaking or fluent in polish language

Exclusion Criteria:

1. Any significant CNS diseases that preceded and not connected with relapse (including seizures, paresis, aphasia, stroke or CNS bleeding, severe brain trauma, dementia, Parkinson's disease, any disease affecting cerebellum, psychosis and diseases involving lack of coordination or movement);
2. Bulky or rapidly progressing disease;
3. Less than 3 months after allo-HSCT transplantation or DLI before screening;
4. The need for high-dose chemotherapy less than 4 weeks before the scheduled apheresis;
5. Concomitant presence of another malignancy and another malignancy diagnosed up to 2 years before inclusion to this trial;
6. Patient's weight below 40 kg and above 130kg
7. Any active bacterial, viral or fungal infection including SARS-CoV2;
8. Latent HBV/HCV/HIV/Syphilis infection;
9. Any other concomitant disease which in the opinion of the investigator would be interfering with the safety of participant in the trial
10. Allergic to penicillin, streptomycin and amphotericin B;
11. Intolerance to cyclophosphamide or fludarabine during previous treatment with these drugs;
12. Chronic systemic immunosuppression treatment (i.e. cyclosporin). Corticosteroids are allowed up to dexamethasone dose of 4 mg a day or equal of this dose;
13. Systemic immunosuppression treatment of acute and/or chronic Graft-versus host disease (GvHD) connected to earlier allogeneic HSCT treatment;
14. Pregnancy;
15. Women in reproductive age as well as men (regardless of age) that do not agree to maintain effective method of contraception during the trial, lactated women can be included into the trial unless declaration of stopping breast feeding during the whole trial time;
16. Unable to provide informed consent for this trial;
17. Lack of actual vaccination against SARS-CoV2 by vaccine accepted to use in the EU;
18. Patients who are not fluent in polish language;
19. Previous use of anti-CD19 CART therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with CRS in particular degree of severity according to ASTCT neurological side effects, febrile neutropenia and infection, cytopenia, other unspecified adverse events and death | through study completion, an average of 1 year
  Safety assessment of IMP administration as the percentage of patients with cytokine release syndrome (CRS) in particular degree of severity according to ASTCT, neurological side effects, febrile neutropenia and infection, cytopenia, other unspecified adverse events and death as a result of the side effects and adverse events described within a 1 month after IMP administration

SECONDARY OUTCOMES:
Percentage of participants with response to the therapy (sum of complete remissions and partial responses in the particular malignancies) | through study completion, an average of 1 year
  Percentage of participants with response to the Tarcidomgen Kimleucel, FCTX-CL19-1 therapy ( best overall response rate defined as the sum of complete remissions and partial responses in the particular malignancies) during one month (1 months, 30 days), three months (3 months, 90 days), twelve months (12 months, 360 days) after IMP administration
Percentage of participants with no possibility to receive the product due to the production failure | through study completion, an average of 1 year
  Percentage of participants with no possibility to receive FCTX-CL19-1 (Tarcidomgen Kimleucel) product that meets the assumed quality criteria due to the production failure

CONTACTS AND LOCATIONS:
Overall Officials: Emilian Snarski, Study Director — FamiCordTx S.A.
Locations (2):
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego - Centralny Szpital Kliniczny, Warsaw, Ul. Banacha 1a
  - Uniwersyteckie Centrum Kliniczne Gdańskiego Uniwersytetu Medycznego - Katedra i Klinika Hematologii i Transplantologii, Gdansk, Ul. Smoluchowskiego 17